CLINICAL TRIAL: NCT06510790
Title: Risk Factors for Bacterial Stent Colonization in Patients With a Double J Ureteral Stent: a Prospective Study
Brief Title: Risk Factors for Bacterial Stent Colonization in Patients With a Double J Ureteral Stent
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ishwor Thapaliya, Prinicpal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 510 (6-11)
Record Dates: First submitted 2024-07-12; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Bacterial Colonization in Double J Ureteral Stent
Keywords: Colonization; Double J stent; Risk factors; Urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — The retained biospecimens are the tips of both the renal and bladder ends of the double J ureteral stent. These tips are cut with a surgical blade and collected in a sterile plastic screw-capped container. They are then sent for bacterial culture and sensitivity testing to identify and evaluate the microorganisms present on the stent. The DNA of these microorganisms can be extracted and analyzed as part of the bacterial evaluation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing DJ stent: All patients coming to TUTH OPD and ER for urological surgery were assessed for the placement of a DJS (polyurethane). Patients fulfilling inclusion criteria were admitted and underwent DJS placement after their respective procedures
  Interventions: Device: Double J stent

INTERVENTIONS:
Device: Double J stent — Double J ureteral catheter has been used to prevent upper urinary tract obstructions or strictures and to facilitate stone clearance after procedures such as percutaneous nephrolithotomy (PCNL), retrograde intrarenal surgery (RIRS), and ureteroscopic lithotripsy (URSL).
  Other Names: Ureteral stent

SUMMARY:
The goal of this prospective study is to identify the risk factors associated with bacterial colonization of DJS and report the common microorganisms isolated and drug susceptibility pattern.

DETAILED DESCRIPTION:
This was a hospital-based prospective observational study performed at a tertiary academic center from March 2022 to August 2023.

All patients coming to TUTH OPD and ER for urological surgery were assessed for the placement of a DJS (polyurethane). Patients fulfilling inclusion criteria were admitted and underwent DJS placement after their respective procedures. All patients received prophylactic antibiotic therapy with levofloxacin for 2 to 3 days at the time of DJS insertion. The DJS was in situ until the duration allocated according to the procedure. The DJS was removed in 2 weeks postoperatively with aseptic precaution under local anesthesia (2% lignocaine jelly) with the help of a 30-degree Karl Storze scope with cystoscope sheath 19/21 and alligator forceps following the standard technique. The equipment was sterilized with a 2.45% Cidex solution for 12 minutes prior to all DJS removal. Then the patient was positioned in the lithotomy position, with proper cleaning of the external genitalia with povidone-iodine 10%, complete separation of the labia in the female, and proper cleaning of the prepuce and glans in the male. Then sterile xylocaine jelly 2% was instilled in the urethra, a cystoscope was inserted into the bladder, alligator forceps were inserted, and a DJS was removed. After removal of the DJS with sterile technique, the tips of both ends (renal end and bladder end) of the stent were cut with surgical blade number 10 and collected in a plastic screw-capped container, and sent for bacterial evaluation.

The report of the culture and sensitivity pattern were collected and treated according to the sensitivity pattern with appropriate antibiotics correlating with the symptoms. Colonization is defined as the growth of microorganisms in the tip culture of either end or both ends of DJS. All the demographic data with other study variables were recorded in proforma. Any amount of preoperative urine albumin from trace amounts and above (+,++, etc.) was considered in this study.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing DJ stent placement

Exclusion Criteria:

* Positive urine culture before stenting
* Taking antibiotics during DJS removal
* Presence of yeasts in urine culture
* Declining informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients coming to TUTH OPD and ER for urological surgery were assessed for the placement of a DJS (polyurethane). Patients fulfilling inclusion criteria were admitted and underwent DJS placement after their respective procedures. All patients received prophylactic antibiotic therapy with levofloxacin for 2 to 3 days at the time of DJS insertion. The DJS was in situ until the duration allocated according to the procedure. The DJS was removed in 2 weeks postoperatively.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Risk factors associated with bacterial colonization of DJS. | 4 weeks
  Patients fulfilling inclusion criteria were admitted and underwent DJS placement after their respective procedures.

SECONDARY OUTCOMES:
The common microorganisms isolated from DJS in culture along with their drug susceptibility pattern. | 4 weeks
  After removal of the DJS with sterile technique, the tips of both ends (renal end and bladder end) of the stent were cut with surgical blade number 10 and collected in a plastic screw-capped container, and sent for bacterial evaluation. The report of the culture and sensitivity pattern were collected and treated according to the sensitivity pattern with appropriate antibiotics correlating with the symptoms. Any amount of preoperative urine albumin from trace amounts and above (+,++, etc.) was considered in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medicine, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The Individual Participant Data (IPD) to be shared for registration on ClinicalTrials.gov will include demographic details (age, sex), preoperative characteristics (hemoglobin levels, albuminuria), procedural information (stent type, duration), microbiological findings (bacterial species, drug sensitivity), and clinical outcomes (complications, mortality). These data will facilitate analysis of risk factors for bacterial colonization in patients with double J ureteral stents and guide future research and clinical practice.
Supporting Information: Study Protocol
Time Frame: Data will be made available after publication of manuscript in the journal.
Access Criteria: Researchers must provide a clear scientific rationale for requesting the data. Data will be shared upon reasonable request to the corresponding author. Requests must detail the intended use of the data and ensure it aligns with the ethical guidelines, ensuring patient confidentiality.